CLINICAL TRIAL: NCT06295757
Title: Effects of Relighting on Smoke Toxicant Deliveries and Subjective Smoking Measures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023LS102; R01CA260831 (NIH)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Tobacco Use; Cigarette Smoking; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking; Tobacco Use Disorder | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Smoking (Other): During the study visits, measures will be taken before and after participants smoke their own usual brand cigarette one continuously. Participants will be randomly assigned to continuous smoking or relight smoking conditions. Participants randomized to the continuous smoking condition will crossover to the relight smoking condition after 60 minutes on their first visit.
  Visits will be separated by 7-10 days, to ensure there are 2 weekdays and 1 weekend day falling in that period for cigarette butt collection.
  On the second visit, participants will begin with the second smoking condition they were assigned on their first visit. They will crossover to the remaining condition after 60 minutes. Participants initially assigned to the continuous smoking condition will begin their second visit with the relighting smoking condition and cross over to the continuous smoking condition after the 60 minutes.
  Interventions: Other: Cigarettes
- Relight Smoking (Other): During the study visits, measures will be taken before and after participants smoke their own usual brand cigarette one continuously. Participants will be randomly assigned to continuous smoking or relight smoking conditions. Participants randomized to the relight smoking condition will crossover to the continuous smoking condition after 60 minutes on their first visit.
  Visits will be separated by 7-10 days, to ensure there are 2 weekdays and 1 weekend day falling in that period for cigarette butt collection.
  On the second visit, participants will begin with the second smoking condition they were assigned on their first visit. They will crossover to the remaining condition after 60 minutes. Participants initially assigned to the relighting smoking condition will begin their second visit with the continuous smoking condition and cross over to the relighting smoking condition after the 60 minutes.
  Interventions: Other: Cigarettes

INTERVENTIONS:
Other: Cigarettes — Participants will smoke their own usual brand cigarettes. Cigarette butts will be collected.

SUMMARY:
Characterize effects of relighting on smoke toxicant deliveries and subjective smoking measures. This will be a within-subject comparison in a single experimental group of 30 smokers who report engaging in relighting behaviors. We will assess smoking intensity for relit and non-relit (i.e., smoked continuously without relighting) cigarettes in the natural environment and will conduct in-clinic measurements of smoking topography and subjective responses for relit and non-relit cigarettes. Information on relighting patterns and smoking topography collected from each participant will be used to compare machine-measured smoke yields of key harmful constituents when their usual cigarettes are smoked with and without relighting. Hypothesis: Relit cigarettes will produce higher levels of toxicants than non-relit cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Smoking at least 10 cigarettes/day for at least 1 year (confirmed by CO > 8 ppm or NicAlert test of 6)
* Engaging in relighting for at least half of their CPD
* No smoking quit attempts in the past month nor intentions to quit in the next month
* Stable medical or psychiatric conditions with systolic blood pressure < 160, diastolic blood pressure < 100 and heart rate < 105 bpm

Exclusion Criteria:

* Participant with current or recent alcohol or drug abuse problems, use of substances of abuse (other than marijuana due to high prevalence of co-use) within the past month
* Currently trying or planning to quit smoking in the next month
* Planning to become pregnant, pregnant or breastfeeding. Pregnancy exclusion will be confirmed through a urine test.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Average Nicotine Level | 1 month
  Level of nicotine in cigarette butts collected during study.

SECONDARY OUTCOMES:
Average Puff Volume | 1 month
  In-clinic measurement of puff volume using topography device.

CONTACTS AND LOCATIONS:
Locations (1):
- Irina Stepanov, PhD, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No